CLINICAL TRIAL: NCT05532020
Title: An Open-Label Study to Assess the Preliminary Efficacy and Safety of DCCR (Diazoxide Choline) Extended-Release Tablets in Patients With Genetic Obesities
Brief Title: An Open-Label Study of Diazoxide Choline in Patients With Genetic Obesities
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soleno Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C615
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: SH2B1 Deficiency Obesity; Obesity Associated With PCSK1 Mutation (rs6232 Variant); SIM1 Deficiency Obesity
Keywords: SH2B1 deficiency obesity; Obesity associated with PCSK1 mutation; (rs6232 variant); SIM1 deficiency obesity; Genetic obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label DCCR (Experimental): 75 - 525 mg DCCR
  Interventions: Drug: DCCR (diazoxide choline) extended-release tablets

INTERVENTIONS:
Drug: DCCR (diazoxide choline) extended-release tablets — All participants will be titrated over a four week period to the maintenance dose. Participants will take DCCR daily for up to 52 weeks.
  Other Names: DCCR

SUMMARY:
This is a phase 2 open-label, one-arm, clinical study to evaluate the efficacy and safety of DCCR (diazoxide choline) extended-release tablets over 1 year of treatment, in patients with genetic obesities.

DETAILED DESCRIPTION:
Patients aged 5 years and older with obesity due to SH2B1 deficiency obesity, obesity associated with PCSK1 mutation (rs6232 variant), or SIM1 deficiency obesity will be enrolled into this phase 2 open-label clinical trial at a single clinical center in North America. All eligible participants will receive DCCR (diazoxide choline) extended-release tablets for 1 year.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide voluntary, written informed consent (parent(s) / legal guardian(s) of patient); provide voluntary, written assent (patients, as appropriate)
* Genetically-confirmed diagnosis of SH2B1 deficiency obesity, obesity associated with PCSK1 mutation (rs6232 variant), or SIM1 deficiency obesity

Key Exclusion Criteria:

* Have participated in an interventional clinical study (i.e., investigational drug or device, approved drugs or device evaluated for unapproved use) within 60 days prior to Screening
* Any known disease and/or condition, which would prevent, in the opinion of the Investigator, the patient from completing all study visits and assessments required by the protocol
* Positive urine pregnancy test (in females of child-bearing potential) or females who are pregnant or breastfeeding, and/or plan to become pregnant or to breast-feed during or within 30 days after study participation

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve at least 5% body weight reduction | Baseline to Week 26
  Proportion of participants who achieve at least 5% body weight reduction

SECONDARY OUTCOMES:
Leptin | Baseline to Week 26
  Change from Baseline in serum leptin
Fasting serum insulin | Baseline to Week 26
  Change in fasting serum insulin
Body fat mass | Baseline to Week 26
  Change in body fat mass (DXA)
Feelings of hunger | Baseline to Week 26
  Change in self-reported feelings of hunger measured on a visual analog scale (VAS), 0 - 100 with 0 being no feelings of hunger and 100 being the most extreme sensation of hunger

IPD SHARING:
Plan to Share IPD: No